CLINICAL TRIAL: NCT03161639
Title: Influence of Working Length Methods in the Performance of Pulpectomies in Primary Teeth - Randomized Clinical Trial
Brief Title: Influence of Working Length Methods in the Performance of Pulpectomies in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Nashalie Andrade de Alencar, Pediatric dentistry PhD student, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Universidade Federal SC
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Endodontically Treated Teeth
Keywords: Pulpectomy; Primary teeth; Working length; Apex locator
MeSH Terms: conditions — Tooth, Nonvital | interventions — Pulpectomy

STUDY DESIGN:
Intervention Model Description: Patients between 6 and 9 years old who search for endodontic treatment in primary teeth. The allocation of subjects to groups will be achieved by randomization. These patients will be randomly divided into 2 groups: G1 - pulpectomy with length measurement performed through radiography and G2 - pulpectomy with length measurement performed with the aid of an apex locator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At the end of the canal access, the first operator will leave the surroundings and a second operator will continue. A length measurement will be determined in order to define the working length. After the working measurement length performed by the second operator, the first operator will be informed about the working length of each canal without the knowledge of which method was used for the length measurement . From then on, the first operator will continue the endodontic treatment. A third operator will evaluate the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Operator 1 (No Intervention): Perform the pulpectomies except the working length measurement
- Operator 2 (No Intervention): Perform the electronic length measurement of the pulpectomies
- Operator 3 (Active Comparator): Perform radiographic length measurement and final evaluation of the pulpectomies
  Interventions: Other: Pulpectomies

INTERVENTIONS:
Other: Pulpectomies — Primary teeth pulpectomy is an important treatment option for necrotic teeth. The correct working length will determine a better chemical and mechanical disinfection of the root canals, without demanding the surrounding periapical tissues and dental germs. In addition, it decreases the chance of a sub or over-filling, which also may interfere with the achievement of the success.
  Arms: Operator 3

SUMMARY:
Verify, through a randomized double-blinded clinical trial, the influence in the performance of pulpectomies in primary teeth, based on two working length methods, electronic and radiographic.

DETAILED DESCRIPTION:
Samples will be composed of children between 6 and 9 years of age, with the need for endodontic treatment in primary teeth. They will be submitted to anamnesis, clinical and radiographic exams for identification of eligibility criteria for the study. These patients will be divided randomly into 2 groups: G1 - pulpectomy with working length method performed through radiography (n=100) and G2 - pulpectomy with working length method performed with the aid of an apex locator (n=100). Endodontic treatment will be done by a single trained operator. After definite restoration and final radiography, an evaluation of the obturation quality will be performed by another blinded operator, who will evaluate the appropriate obturation length. The clinical treatment success and the radiographies will also be analyzed during a period of 24 months through clinical and radiographic exams, also by a blinded operator.

ELIGIBILITY:
Inclusion Criteria:

* Primary molars teeth with caries or defected restorations associated with signs or symptoms of irreversible pulpal inflammation - spontaneous pain or pulpal necrosis - presence of abscess, fistula, edema, periapical or inter-radicular radiolucency

Exclusion Criteria:

* Primary molars teeth previously manipulated, with obliteration of the root canal, with bone reabsorption involving the crypt of the permanent tooth, internal or external pathological or physiological reabsorption involving more then half of the shortest root and unrestorable tooth

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2020-09-02 (Estimated)

PRIMARY OUTCOMES:
Outcome Electronic Apex locator | Evaluations will be done during 24 mouths after the pulpectomy performance
  The use of an electronic apex locator for the achievement of working length in primary teeth pulpectomies will demonstrate a similar or better result than the radiographic method for the obturation adequacy. Also it will show a closer or a better result in the evaluation of the clinical and radiographic success in a long-term treatment.

SECONDARY OUTCOMES:
Difference in length measurement methods for pulpectomies in primary teeth | Evaluations will be done during the pulpectomy performance
  Evaluate if there is a significant difference in the accuracy of electronic apex locators compared to the conventional radiography in working length measurements
Influence of working length measurement methods in the obturation level of pulpectomy in primary teeth | Evaluations will be done after the pulpectomy performance
  Evaluate the effect of two working length measurement methods in the obturation level of pulpectomy in primary teeth

CONTACTS AND LOCATIONS:
Overall Officials: Nashalie Alencar, Ms, Principal Investigator — Universidade Federal de Santa Catarina
Locations (2):
- Brazil (2):
  - Nashalie Andrade de Alencar, Florianópolis, Santa Catarina
  - Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ravanshad S, Adl A, Anvar J. Effect of working length measurement by electronic apex locator or radiography on the adequacy of final working length: a randomized clinical trial. J Endod. 2010 Nov;36(11):1753-6. doi: 10.1016/j.joen.2010.08.017. Epub 2010 Sep 19. PMID 20951282